CLINICAL TRIAL: NCT04237402
Title: Demonstration of the Presence of a Carbonyl Stress in the Hair Follicles of Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STRESSCARBONYL2
Record Dates: First submitted 2019-10-01; First posted 2020-01-23 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Telogen Effluvium

STUDY DESIGN:
Intervention Model Description: 2 sampling timepoints:
  * before delivery
  * after delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra individual (Other): Before and after pregnancy, hair follicles will be analysed
  Interventions: Other: Hair follicles sampling

INTERVENTIONS:
Other: Hair follicles sampling — The hair follicles will be collected by strand of 5 to 6 hairs approximately in the scalp (centro-parietal part), in order to obtain 20 follicles with epithelial sheath.

SUMMARY:
In this study, the investigator will try to highlight the presence of carbonyl compounds in the hair follicles of postpartum women by comparing these compounds before and after delivery.

DETAILED DESCRIPTION:
At the cutaneous level, oxidative stress induces the formation of carbonyl compounds which, by binding to proteins, produce non-functional adducts inducing cutaneous aging. This mechanism is called "carbonyl stress".

During pregnancy, estrogen increases massively, stimulates the whole body and prolongs the life of the hair (slower passage in telogen phase).

After delivery, estrogen levels drop, resulting in a massive and simultaneous hair loss that should have "naturally" fallen earlier. In addition, birth is a stressful stage for most moms. This stress and excessive fatigue and possibly a return to work may also be responsible for hair loss.

Is the carbonyl stress also present in the scalp and can it be one of the mechanisms involved in the occurrence of postpartum hair loss? To demonstrate this, samples of hair follicles are taken. The proteins are extracted from the samples and then assayed. The oxidized (carbonyl) proteins are labeled with specific fluorescent probes

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the Population:

* Pregnant woman (≥ 33 weeks of amenorrhea)
* Woman aged between 18 and 40 years (included)
* Phototype I to IV included according to Fitzpatrick's classification
* Affiliation to a French social security scheme or benefiting from such a scheme
* Signed informed consent form

Exclusion Criteria:

Criteria related to the Population:

* High risk or pathological pregnancy, according to the opinion of the investigator
* Deprivation of liberty by administrative or judicial decision or subject under guardianship
* Impossibility, according to the investigator, to comply with the requirements of the protocol
* Linguistic or psychic incapacity to sign informed consent
* Concomitant participation in a clinical study that may interfere with the results of the study, according to the opinion of the investigator (excluding observational studies)

Criteria related to Pathology :

* Alopecia causing hair loss on the upper part of the scalp
* Dermatological pathology or evolving cutaneous lesion in the scalp
* Known history of hepatitis B and C, HIV
* Past or present neoplastic condition
* Acute evolving pathology
* Gestational diabetes treated with insulin

Criteria related to Treatments:

* Treatment of general thyroid disorders initiated or modified for less than 3 months prior to inclusion (or change of specialty for less than 3 months)
* Systemic treatment affecting hair growth taken for at least 4 weeks during the 3 months prior to inclusion
* Systemic treatment: nonsteroidal anti-inflammatory drug, corticosteroid, antibiotic, antihistamine taken for 5 consecutive days within 2 weeks prior to inclusion or that may interfere with the results of the study according to the investigator,
* Dermal use, for at least 4 weeks, of Minoxidil, Aminexil within 3 months prior to inclusion
* Dermal use in the 4 weeks prior to inclusion, of any product that may be active on the hair follicle and scalp or may affect the dosage of carbonyl compounds (including hair dyes)
* Last shampoo less than 2 days before the inclusion and application of styling / care products (gel, lacquer, wax, conditioner ...) or water between the last shampoo and the inclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 20 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Change of biological evaluation | 1st sample: inclusion visit (up to 8 weeks before delivery)- 2nd sample: end of study visit (10 to 16 weeks after delivery)
  Evaluation of the quantity of carbonyl compounds measured in the hair follicles taken before and after delivery.

SECONDARY OUTCOMES:
Safety evaluation | From inclusion to end of study
  Adverse events evaluation for all subjects, all along the study

CONTACTS AND LOCATIONS:
Overall Officials: Christophe VAYSSIERE, MD, Principal Investigator
Locations (1):
- Hôpital Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No
Proof of concept study, with confidential data